CLINICAL TRIAL: NCT04765371
Title: Comparison Between Prednisolone and Dexamethasone on D28 Mortality in Patients on Oxygen Therapy, with CoViD-19: Multicenter, Randomized, Open-label Non-inferiority Study
Brief Title: Comparison Between Prednisolone and Dexamethasone on Mortality in Patients on Oxygen Therapy, with CoViD-19
Acronym: COPreDex
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRD1520; 2020-005883-78 (EudraCT Number)
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-05

CONDITIONS: Coronavirus Infection
Keywords: Coronavirus Infections; SARS-CoV-2; Corticostéroïdes; Severe form of COVID-19
MeSH Terms: conditions — Coronavirus Infections | interventions — Dexamethasone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEXAMETHASONE Arm (Active Comparator): Patients will take 6 mg per day of Dexamethasone during 10 days
  Interventions: Drug: DEXAMETHASONE
- PREDNISOLONE Arm (Active Comparator): Patients will take 60 mg per day of Prednisolone during 10 days
  Interventions: Drug: PREDNISOLONE

INTERVENTIONS:
Drug: DEXAMETHASONE — Patients will take 60 mg per day of Prednisolone (40 mg morning and 20 md evening) between D1 to D10
  Other Names: DEXAMETHASONE Arm
  Arms: DEXAMETHASONE Arm
Drug: PREDNISOLONE — Patients will take 60 mg per day of Prednisolone (40 mg morning and 20 md evening) between D1 to D10
  Other Names: PREDNISOLONE Arm
  Arms: PREDNISOLONE Arm

SUMMARY:
The aim of the study is to evaluate two differents regimens of corticosteroids (prednisolone versus dexamethasone) on D28 mortality in patients with CoViD 19 pneumonia requiring oxygen supplementation

DETAILED DESCRIPTION:
Low-dose glucocorticoid treatment is the only medication showing a significant reduction in mortality in cases of COVID-19 pneumonia requiring oxygen supplementation or ventilatory support.

Intravenous or oral dexamethasone are well evaluated in randomized study but other oral corticosteroids are not. Compared to dexamethasone, prednisolone is more available in France and easily taken by patients, especially in case of home medical care.

The pharmacokinetics/pharmacodynamics of prednisolone and dexamethasone are different. To obtain similar effects, prednisolone should be theoretically taken twice a day and at a superior dose than the strict prednisone equivalence of 6mg dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient with SARS-CoV-2 pneumopathy documented by nasopharyngeal or bronchoalveolar lavage fluid RT-PCR or any documented clinical symptoms support by CT scan
* Patient with SpaO2 ≤ 94 % in room air (90% for patient with respiratory failure) and requiring an oxygen therapy
* Negative pregnancy test for women of childbearing age
* Informed and written informed consent (IC) obtained
* Patients with affiliation to the social security system

Exclusion Criteria:

* Patient with corticosteroids as background treatment (≥ 10 mg equivalent)
* Patient under supplemental oxygen > 6 L/min
* Immunocompromised patient (AIDS, bone marrow or solid organ transplants, etc.)
* Patient who received a corticosteroid dose within 3 days for Covid-19
* Medical history of hypersensitivity to Prednisolone or Dexamethasone; or lactose / galactose (excipients with known effect)
* Another active virus such hepatitis, herpes, varicella, shingles ….
* Psychotic state not controlled by treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Mortality assessment at D28 | At Day 28
  Assessment of vital status at D28 in Dexamethason arms vs Prednisolone arms

SECONDARY OUTCOMES:
Assessment of clinical course in both groups (arms) | At Day 28
  The clinical course for each patient will be measured, for several items, and compared between both groups to see if a significant difference is observed.
  Items, considered for comparison, are listed below :
  * Number of oxygen therapy days,
  * Number of patients requiring oxygen therapy increase (High-Flow Oxygen Therapy, CPAP/BIPAP, mechanical ventilation, ECMO)
  * Number of hospital days
  * Number of patient admitted in Resuscitation Unit /Intensive care Unit
  * Number of patient with organic damage other than lung
  * Number of disease-related infection other than SARS-Cov-2
  * Frequency and evolution of complication of corticosteroid therapy (Severity evaluated according to CTCAE (diabetes, acute psychosis or other adverse effect consider to be link to corticosteroide therapy by investigator))
Measurement of evolution of respiratory symptoms in both groups (arms) | From Day 0 to Day 28
  Evolution of respiratory symptoms will be measured for each patient, for several items, and compared between both groups to see if a significant difference is observed.
  Items, considered for comparison, are listed below :
  * Oxygen saturation rate,
  * Oxygen flow,
  * Respiratory rate
Assessment of patient satisfaction towards the treatment | At Day 28
  Assessment of patient satisfaction with a satisfaction questionnaire (Likert-type scale) For each item, patient ticks : Very satisfied, Satisfied, Unsatisfied or Very unsatisfied
Comparison betwween D1 and D28 of patient quality of life evolution between randomization groups (arms) | At Day 1 and Day 28
  Measurement of patient quality of life evolution with EQ5D self-assessment questionnaire at day1 and day 28.
  For item of mobility, autonomy and current activities, patient ticks : I have no problem, I have some problems or I am I am unable to do For item of pain and anxiety/depression, patient ticks : no, moderate or severe
Comparison betwween D1 and D28 of adverse events and adverse effects between randomization groups (arms) | At Day 28
  Measurement of adverse events number and adverse effects number during the 28 days of the study

CONTACTS AND LOCATIONS:
Overall Officials: Dr Edouard DEVAUD, Principal Investigator — Hôpital NOVO
Locations (8):
- France (8):
  - Department of Emergency, Hospital Victor Dupouy, Argenteuil
  - Department of Pneumology and Infectious Medicine, Hospital Carnelle Portes de l'Oise, Beaumont
  - Department of Infectious and Tropical Diseases, Hospital Simone Veil, Eaubonne
  - Department of Infectious Medicine, Hospital of Gonesse, Gonesse
  - Department of Internal Medicine, Hospital Emile Roux - Le Puy-en-Velay, Le Puy-en-Velay
  - Department of Infectious and Tropical Diseases, Hospital René Dubos,, Pontoise
  - Department of Infectious and respiratory Diseases, Hospital Delafontaine, Saint-Denis
  - Department of Pneumology and Infectious Diseases, Hospital of Saint-Quentin, Saint-Quentin

IPD SHARING:
Plan to Share IPD: No